CLINICAL TRIAL: NCT06679894
Title: Evaluation of Implant Stability Changes in Sites Prepared with Different Osseodensification Techniques: a Prospective Observational Clinical Study
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-IND-9
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Edentulous; Alveolar Process Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Single tooth edentulism right: single missed teeth
  Interventions: Procedure: Implant site preparation with osteotomes and electrified mallet
- single tooth edentulism left: single missed tooth
  Interventions: Procedure: Implant site preparation with osseodensification drills

INTERVENTIONS:
Procedure: Implant site preparation with osteotomes and electrified mallet — Under local anesthesia (mepivacaine HCL 2% with epinephrine1:100.000), a minimally invasive full-thickness flap was elevated to expose the alveolar crest.
  A pilot osteotome (100-P) was used to easily perforate the cortical plate. Subsequently, osteotomes with gradually increasing diameters were employed until the final diameter of 3.2 mm was reached.
  The sequence of osteotomes and their respective diameters were as follows:
  1. Osteotome 100-P: At a height of 8.5 mm, the diameter was 2.2 mm;
  2. Osteotome 160: At a height of 8.5 mm, the diameter was 2.8 mm;
  3. Osteotome 200: At a height of 8.5 mm, the diameter was 3.2 mm. Implant (4.0x8.5 mm; Anyridge, Megagen, Gyeongbuk, South Korea) was positioned using a surgical motor.
  A 3 mm high transepithelial abutment (OCTA, Megagen, Gyeongbuk, South Korea) was connected to it using a torque wrench and it was tightened to 30 Ncm.
  Single sutures in monofilament synthetic polypropylene 4.0 were performed to close flaps around the abutment.
  Groups: Single tooth edentulism right
Procedure: Implant site preparation with osseodensification drills — Under local anesthesia (mepivacaine HCL 2% with epinephrine1:100.000), a minimally invasive full-thickness flap was elevated to expose the alveolar crest.
  The implant site preparation was realized using osseodensification burs at a rotation speed of 1200 rpm. The osseodensification burs sequence was as follows:
  1. Initial pilot hole (rotated clockwise);
  2. WT1828 bur (rotated counterclockwise),
  3. WT2838 bur (rotated counterclockwise). Implant (4.0x8.5 mm; Anyridge, Megagen, Gyeongbuk, South Korea) was positioned using a surgical motor.
  A 3 mm high transepithelial abutment (OCTA, Megagen, Gyeongbuk, South Korea) was connected to it using a torque wrench and it was tightened to 30 Ncm.
  Single sutures in monofilament synthetic polypropylene 4.0 were performed to close flaps around the abutment.
  Groups: single tooth edentulism left

SUMMARY:
The goal of this observational study is to compare, within a cohort of patients requiring rehabilitation in two different sites of the premolar area in the upper maxilla, the primary and secondary stability of implants placed in sites prepared using a magnetic mallet and osseodensification burs.

DETAILED DESCRIPTION:
The primary outcome measures included implant primary stability, assessed through insertion torque and ISQ (Implant Stability Quotient).

Secondary outcome measures were implant secondary stability pattern during the initial 90 days post-implant placement (ISQ), implant survival after one year, the time required for each implant site preparation and any complications or adverse events.

As an additional outcome of this study, we aimed to assess whether there was a relationship between the instrument utilized for implant site preparation and early marginal bone loss. Marginal bone levels were measured at three time points: immediately after surgery (T0), upon delivery of prosthetic rehabilitation (T1), and after one year of loading (T2). The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.

Study design: Observational study of a prospective non-profit cohort.

Study population: The study will be conducted in an outpatient hospital setting.

Sample size calculation: Data from the literature were used regarding insertion torque with the use of the magnetic mallet and osseodensification burs. On average, these data ranged from 50 to 70 Ncm for the magnetic mallet and 35 to 59 Ncm for the osseodensification burs. Using a statistical power of 80%, an alpha error of 0.05, and a beta error of 0.2, the sample size was calculated to be six patients for the experimental group (magnetic mallet - MM) and six patients for the control group (osseodensification burs - OD).

Enrollment procedure: All patients who meet the inclusion and exclusion criteria will be enrolled in the study following the administration of the Information Sheet and the acquisition of informed consent.

Patients seeking implant-supported rehabilitation due to the absence of at least two teeth were evaluated with a periapical radiograph at each selected site to assess the adequacy of residual bone height. If the available bone height appeared to be sufficient, a second-level radiographic exam, a Cone Beam Computed Tomography (CBCT), was performed to evaluate whether the bone volume was adequate for supporting implant rehabilitation.

Surgical phase: After performing local anaesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap was elevated. The surgeon, who conducted all the procedures, initiated the first implant site preparation using osteotomes and electrified mallet (Magnetic Mallet, Metaergonomica, Milan, Italy) (test group).

Meanwhile, a second operator began timing the duration of surgery from the initial bone contact of the first osteotome to the placement of the implant.

All the procedures strictly followed the manufacturer's recommendations: initially, a pilot osteotome (100-P) was used. Osteotomes with gradually increasing diameters were employed until the final diameter of 3.2 mm was reached. Subsequently, a 3 mm high transepithelial abutment (OCTA, Megagen, Gyeongbuk, South Korea) was connected to it using a torque wrench and it was tightened to 30 Ncm. Single sutures in monofilament synthetic polypropylene 4.0 were performed to close flaps around the abutment.

Right after the suture of the first surgical site, the site preparation of the control group began.

After performing local anaesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap was elevated; the surgeon initiated the preparation using osseodensification burs (Densah, Versah, Jackson, USA). Another operator started timing at the beginning of the procedure and concluded when the implant was placed in the final position.

The experimental sites were prepared using osseodensification burs (Densah, Versah) at a rotation speed of 1200 rpm. The implant beds were equal in dimension and diameter to those prepared with the magnetic hammer, 8.5 mm in height and 3.2 mm in diameter. Subsequently, a 3 mm high transepithelial abutment (OCTA, Megagen, Gyeongbuk, South Korea) was connected to it using a torque wrench and it was tightened to 30 Ncm. Single sutures in monofilament synthetic polypropylene 4.0 were performed to close flaps around the abutment.

After surgery, a radiographic control was conducted to evaluate the correct positioning of the implants.

Once completed, a blinded operator measured ISQ values of each implant from two different directions: vestibular-palatal and mesio-distal.

Each measurement was taken at abutment level three times for each direction, and their averages were used for the statistical analysis.

The values were collected using a Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg # 74, Osstell, Göteborg, Sweden).

After surgery, a check-up visit was scheduled after one week, when the sutures were removed, soft tissue healing was evaluated, and ISQ was measured as in the first time.

The subsequent check-ups were scheduled at 14 days, 21 days, 28 days, 60 days, 90 days and in each meeting, the same parameters were re-evaluated.

All the implants were restored with screw-retained single metal-ceramic crowns four months after surgery and then followed up for at least for 12 months after prosthetic loading. Two additional check-ups were scheduled for radiographic control after 6 months and 1 year.

Statistical plan: The statistical analysis will be performed by means of a computerized statistical package (SigmaStat 3.5, SPSS Inc., Germany). The data will be expressed as mean ± standard deviation and median (interquartile range), respectively, for parametric and non-parametric values.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old;
* Indication for an implant-supported rehabilitation in the upper premolar / first molar areas;
* The area in which the implants will be placed must have had at least 6 months of healing;
* No use of grafts or bone substitutes following tooth extraction;
* Bone volume measuring at least 10 mm in height and 6 mm in width;
* In case of two adjacent implants the distance between the natural teeth must be at least 14 mm, composed by twice the width of each implant (4 mm), the distance between them (at least 3 mm) and twice the distance between each teeth (at least 1,5 mm)
* Bone quality belonging to class D3 or D4, following Misch classification
* Absence or decision to not wear a removable prosthesis during the healing period;
* Patients with good and stable oral hygiene;
* Signed informed consent form.

Exclusion Criteria:

* Acute myocardial infarction within the previous six months;
* Uncontrolled bleeding disorders;
* Uncontrolled diabetes (HBA1c > 7.5%);
* Radiotherapy in the head-neck area in the previous 48 months;
* Immunocompromised patients (es. AIDS / chemotherapy);
* Current or previous treatment with antiresorptive drugs via intravenous injection;
* Psychological or psychiatric disease;
* Alcohol and /or drugs abuse;
* Heavy smokers (more than 10 cigarettes / day);
* Plaque index >20% and/or bleeding on probing >10%
* Pregnant or breastfeeding patients;
* Patients refusing to participate in follow-up checks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After investigating general and local anamnesis, which included evaluation of systemic illnesses and potential allergies, a dental visit was conducted to formulate a specific treatment plan.
  If the patient was deemed eligible for the research protocol, an additional periapical radiograph was obtained for each selected site to assess the adequacy of residual bone height.
  If the available bone height appeared to be sufficient, a second-level radiographic exam, a Cone Beam Computed Tomography (CBCT), was performed to evaluate whether the bone volume was adequate for supporting implant rehabilitation.
  For patients requiring tooth extraction, this second assessment was performed after six months of healing after extraction.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Implant primary stability | At implant insertion
  Insertion torque
Implant primary stability | At implant insertion
  Resonance frequency

SECONDARY OUTCOMES:
Implant secondary stability | 7 days after implant insertion
  Resonance frequency
Implant secondary stability | 14 days after implant insertion
  Resonance frequency
Implant secondary stability | 21 days after implant insertion
  Resonance frequency
Implant secondary stability | 28 days after implant insertion
  Resonance frequency
Implant secondary stability | 60 days after implant insertion
  Resonance frequency
Implant secondary stability | 90 days after implant insertion
  Resonance frequency
Surgical time | The measurement began when the first pilot osteotome or drill was used and ended when the implant was placed.
  In seconds

OTHER OUTCOMES:
Peri-implant marginal bone level stability | Immediately after surgery
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.
Peri-implant marginal bone level stability | Upon delivery of prosthetic rehabilitation (6 months after surgery)
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.
Peri-implant marginal bone level stability | One year of loading
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Piezosurgery Academy, Parma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No